CLINICAL TRIAL: NCT06887465
Title: Comparison of Non-Invasive Wearable Sensors to Radial Arterial Catheterization on Human Subjects
Brief Title: Non-invasive and Continuous Blood Pressure Monitoring
Status: Not yet recruiting | Type: Observational
Sponsor: Vena Vitals (Industry)
Collaborators: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: VVAL0001
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Blood Pressure
Keywords: Blood pressure monitoring; Non-invasive Blood Pressure Monitoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Non-invasive Blood Pressure Monitor — Application of the VeriTrack non-invasive blood pressure monitor

SUMMARY:
The goal of this observational study is to evaluate the accuracy and reliability of the VeriTrack non-invasive blood pressure monitor compared to radial arterial catheterization in adult surgical patients.

The main question it aims to answer is:

How well does VeriTrack measure continuous blood pressure compared to an arterial catheter?

Researchers will compare VeriTrack readings to arterial line measurements to determine if the VeriTrack provides comparable accuracy and clinical utility.

Participants will wear the VeriTrack device during surgery and have a radial arterial catheter placed as part of standard care.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose blood pressure will be monitored using an arterial line during their procedure
* Patients who have a palpable dorsalis pedis pulse

Exclusion Criteria:

* Patients who have non-palpable dorsalis pedis pulses
* Patients whose limbs are inaccessible for placement of Vena Vitals Wearable
* Patients with known allergy to adhesives and/or silicone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery who have an arterial line and are in supine position
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the VeriTrack device in continuous blood pressure monitoring | 1-24 hours
  Systolic, diastolic, and mean arterial pressure (MAP) values will be compared between the VeriTrack and the arterial line using a Bland-Altman analysis.

SECONDARY OUTCOMES:
Blood Pressure Change Accuracy | 1-24 hours
  Changes in sys, dia, and MAP measured by VeriTrack will be evaluated and compared to the changes measured by the arterial line

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided